CLINICAL TRIAL: NCT07209995
Title: Ultrasound Guided Retroclavicular Infraclavicular Versus Axillary Block as Regional Anesthesia in Obese Patients Undergoing Around and Below Elbow Surgeries: A Randomized Clinical Study
Brief Title: Ultrasound Guided Retroclavicular Infraclavicular Versus Axillary Block as Regional Anesthesia in Obese Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#1680/23-Sep-2025
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Achievement of High-quality Analgesia in Elbow Surgeries
Keywords: retroclavicular infraclavicular approach the axillary block obese patients elbow surgeries.

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (R) (Active Comparator): Patients will recieve retroclavicular infraclavicular brachial plexus block
  Interventions: Other: retroclavicular infraclavicular brachial plexus block for
- Group (A) (Active Comparator): Patients will receive the axillary brachial plexus
  Interventions: Other: axillary block

INTERVENTIONS:
Other: retroclavicular infraclavicular brachial plexus block for — The patient will be placed supine, head facing the contralateral side. A high- frequency 13-6 MHz linear array transducer probe will be placed medial to the coracoid process below and perpendicular to the clavicle to obtain a short-axis view of the cords of the brachial plexus and the axillary vessels. The needle will be inserted in the supraclavicular fossa, approximately one cm posteriorly to the clavicle, and advanced in plane parallel to the probe. After passing the initial blind zone of about 2 cm caused by the clavicle's acoustic shadow, the needle tip will be continuously seen, until it appears posterior to the axillary artery. A single injection of the local an esthetic will be performed without needle repositioning unless paresthesia is elicited
  Arms: Group (R)
Other: axillary block — The axillary nerve block is performed from behind the patient with the patient seated. The axillary nerve will be identified within the quadrilateral space by placing high frequency linear probe parallel to the long axis of the humeral shaft. The nerve was identified next to the circumflex artery
  Arms: Group (A)

SUMMARY:
The purpose of this study is to compare the analgesic outcomes (time to first analgesic request, total amount of analgesic consumption, and pain scores) following the ultrasound-guided retroclavicular infraclavicular approach and the axillary approach in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients acceptance to share in the study.
* Patients with ASA physical status I-II.
* Obese patients (BMI 30-40 kg/m²) undergoing around and below elbow surgeries under regional anesthesia.
* Patients requiring a single injection infraclavicular retroclavicular brachial plexus block or axillary block for around and below elbow surgeries.

Exclusion Criteria:

* Patients with a history of allergic reactions or contraindications to local anesthetics.
* Patients with significant comorbidities (e.g., severe cardiovascular, neurological, or musculoskeletal disorders).
* Patients with a history of previous shoulder or clavicle surgery that may distort anatomy and affect the efficacy of the block.
* Pregnant or breastfeeding women.
* Patients with a history of systemic infections or skin infections in the area of the block.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request in each group | 24 hours postoperative

SECONDARY OUTCOMES:
Block assessment and definition of successful block | 30 minutes after the block
Imaging time | the time between probe application and insertion of the needle
Needle time | the time between insertion of the needle and complete injection of local anesthetic
-Procedure time | the summation of the imaging and needling times
Pain intensity | basal, one, 2, 4, 8, 12, 16, 20 and 24 hours postoperative
  10-point NRS [(0 = no pain, 10 = worst imaginable pain), 1 - 3: Mild pain (nagging, annoying, slightly interfering with activities of daily living (ADLs), 4 - 6: Moderate pain (significantly interfering with ADLs, 7 - 10: Severe pain (disabling, unable to perform ADLs)]
Total analgesia need | the first postoperative 24 hours
Duration of the sensory block | first 24 hours postoperative
Duration of the motor block | first 24 hours postoperative
Incidence of block complications | first 24 h0urs postoperative
  hematoma formation or paresthesia or local anesthetic systemic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Howida A Kamal, MD, Study Director — faculty of medicine,zagazig university Egypt
Locations (1):
- faculty of medicine,zagazig university Egypt, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided